CLINICAL TRIAL: NCT01559623
Title: Colonization of the Female Urethra With Mycoplasma Hominis, Ureaplasma Urealyticum, Chlamydia Trachomatis, or Neisseria Gonorrhea in Patients With Lower Urinary Tract Symptoms
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: OAB2012
Record Dates: First submitted 2012-03-19; First posted 2012-03-21 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Overactive Bladder Syndrome

STUDY DESIGN:
Time Perspective: Retrospective

INTERVENTIONS:
Procedure: retrospective data analysis — retrospective data analysis

SUMMARY:
The purpose of this study is to assess the prevalence of mycoplasma hominis, ureaplasma urealyticum, neisseria gonorrhea, and chlamydia trachomatis in women with overactive bladder symptoms, and to correlate these findings with cystoscopic and urodynamic findings.

ELIGIBILITY:
Inclusion criteria:

* women with urogynecologic and urodynamic examination at our institution between 1.1.2009 and 31.12.2011

Exclusion criteria:

* none

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: clinic for urogynecology
Sampling Method: Non-Probability Sample
Enrollment: 766 (Actual)
Dates: Start 2009-01; Primary Completion 2011-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
prevalence of ureaplasma urealyticum | time of urogynecologic assessment
prevalence of mycoplasma hominis | time of urogynecologic assessment
prevalence of neisseria gonorrhea | time of urogynecologic assessment
prevalence of chlamydia trachomatis | time of urogynecologic assessment

CONTACTS AND LOCATIONS:
Overall Officials: David Amos Scheiner, MD, Principal Investigator — University Hospital Zurich, Division of Gynecology
Locations (1):
- University Hospital Zurich, Gynecology, Zurich, Canton of Zurich, Switzerland